CLINICAL TRIAL: NCT02337270
Title: Phase 1, Open-label Clinical Trial to Evaluate the Safety and Immunogenicity of an Adenovirus-based Tuberculosis Vaccine Administered by Aerosol
Brief Title: Phase 1 Clinical Trial of the Safety and Immunogenicity of an Adenovirus-based TB Vaccine Administered by Aerosol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M002
Record Dates: First submitted 2014-12-19; First posted 2015-01-13 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Vaccine; Aerosol; Adenovirus; Immunogenicity
MeSH Terms: conditions — Tuberculosis; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Aerosol (Experimental): Receive 10^6 Ad5Ag85A by aerosol at day 0
  Interventions: Biological: Ad5Ag85A
- Group 2 Aerosol (Experimental): Receive 2x10^6 Ad5Ag85A by aerosol at day 0
  Interventions: Biological: Ad5Ag85A
- Group 3 Intramuscular (Experimental): Receive 10^8 Ad5Ag85A by intramuscular injection at day 0
  Interventions: Biological: Ad5Ag85A

INTERVENTIONS:
Biological: Ad5Ag85A — Aerosol administration of Ad5Ag85A

SUMMARY:
This is a phase 1 study, in healthy volunteers who have previously been immunized with bacilli Calmette Guerin (BCG), to evaluate the safety and immune responses that develop in the blood and lungs following the administration by aerosol of a new experimental adenovirus-based vaccine for tuberculosis (TB), Ad5Ag85A.

DETAILED DESCRIPTION:
This is a phase 1, open label study to evaluate the safety and immunogenicity of a single administration of one of two doses of a recombinant replication deficient human adenoviral (Ad5) TB vaccine containing the immunodominant antigen Ag85A delivered to the respiratory tract by aerosol in healthy volunteers with a history of BCG immunization.

28 healthy volunteers will be enrolled. The first cohort (n=8) will receive a lower dose of vaccine using the AeroNeb Solo Vibrating Mesh Nebulizer. For the second cohort (n=20) participants will be randomized to either a higher dose of vaccine by aerosol (n=10) or intramuscular administration (n=10). Cellular immune responses in the lung and peripheral blood will be evaluated

ELIGIBILITY:
Inclusion Criteria:

1. Healthy human subjects who are between 18 and 55 years of age with a history of BCG vaccination.
2. HIV antibody negative
3. Able to understand and comply with protocol requirements and instructions; able to attend scheduled study visits and complete required investigations.
4. For women, negative pregnancy test and practicing two acceptable forms of contraception for the duration of the study (barrier contraceptive, birth control pill, surgically sterile, post-menopausal 2 years, abstinence)
5. For men, using barrier contraception for the duration of the study

Exclusion Criteria:

1. Pregnant or lactating women
2. Subjects who have any acute or chronic illnesses including active tuberculosis, any relevant findings on physical examination or are receiving any drug treatment in the opinion of the investigator likely to affect the immune system including current use of inhaled or nasal steroids.
3. Subjects with a history of any bleeding disorder or receiving any drug treatment that in the opinion of the investigator may increase the risk of bleeding
4. Subjects with a history of respiratory disease, e.g. asthma, chronic bronchitis, chronic obstructive pulmonary disease (COPD).
5. Current smokers, including e-cigarettes, and ex-smokers who have quit within the last year, as reported by the subject
6. Subjects with clinically significant abnormality of baseline spirometry tests
7. Any health-related condition for which study bronchoscopy is contraindicated
8. Subjects who have a history of active or latent TB infection or whose PBMC's are responsive to ESAT6/CFP10 stimulation using a commercial interferon gamma release assay for TB [consistent with latent TB infection].
9. Subjects whose baseline laboratory values are outside of the normal range unless the abnormality is considered not to be of clinical relevance by the Investigator. A single repeat test is allowed during the screening period.
10. Subjects whose use of alcohol or drugs would, in the opinion of the investigator, interfere with adherence to the study protocol.
11. Subjects who are using, or have a history of using, inhaled cocaine, metamphetamine or other inhaled or smoked recreational drugs. Subjects who give a history of last smoking marijuana more than a year ago may be enrolled, as long as they do not smoke marijuana for the duration of the study.
12. Failure to provide written consent.
13. Known allergy to vaccine components
14. Previous vaccination with Ad5Ag85A or any other experimental TB vaccine
15. Known exposure to active TB within past 6 months or subjects whose occupation puts them at increased risk of TB exposure (based on Hamilton Health Science/St Joseph Healthcare list of high risk personnel)
16. Any abnormality on chest x-ray suggestive of active or remote tuberculosis infection or evidence on chest-x-ray of clinically significant respiratory disease.
17. PPD skin test within last 12 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting adverse events | Over 24 weeks
  Adverse events will be assessed according to the CTCAE Expanded Common Toxicity Criteria at 48-72 hours after vaccination, and at weeks 2, 4, 8, 12, 16 and 24

SECONDARY OUTCOMES:
Immunogenicity of one of two doses of Ad5Ag85A administered by aerosol | Two weeks after vaccination
  Change from baseline in the immune responses of specific T-cells in bronchoalveolar lavage [BAL] fluid (mucosal) and blood (systemic). Immune responses measured will include interferon Elispot assay, cytokine production and intracellular cytokine staining
Immunogenicity of one of two doses of Ad5Ag85A administered by aerosol | Eight (first cohort) or twelve (second cohort) weeks after vaccination
Immunogenicity of inhaled administration of Ad5Ag85A compared with intramuscular administration | Two weeks after vaccination
Immunogenicity of inhaled administration of Ad5Ag85A compared with intramuscular administration | Twelve weeks after vaccination
Number of participants reporting adverse events with inhaled administration of Ad5Ag85A compared with intramuscular administration | Over 24 weeks
Immune responses measured from induced sputum compared with bronchoalveolar lavage | Two weeks after vaccination
  For first cohort of 8 participants only
immune responses measured from induced sputum compared with bronchoalveolar lavage | Eight weeks after vaccination
  For first cohort of 8 participants only
Number of participants developing a positive interferon release assay for TB after vaccination with Ad5Ag85A | At 16 weeks
  For first cohort of 8 patients only
Number of participants reporting adverse events correlated with level of pre-existing anti-adenoviral antibodies | Over 24 weeks
Immune response to vaccination correlated with pre-existing anti-adenoviral antibodies | Two weeks after vaccination
Immune response to vaccination correlated with pre-existing anti-adenoviral antibodies | Eight weeks after vaccination
Number of participants reporting adverse effects correlated with dose of vaccine received by inhalation | Over 24 weeks
Immune response to vaccine correlated with dose of vaccine received by inhalation | Two weeks after vaccination
Immune response to vaccine correlated with dose of vaccine received by inhalation | Eight or 12 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Fiona M Smaill, MB,ChB, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Jeyanathan M, Fritz DK, Afkhami S, Aguirre E, Howie KJ, Zganiacz A, Dvorkin-Gheva A, Thompson MR, Silver RF, Cusack RP, Lichty BD, O'Byrne PM, Kolb M, Medina MFC, Dolovich MB, Satia I, Gauvreau GM, Xing Z, Smaill F. Aerosol delivery, but not intramuscular injection, of adenovirus-vectored tuberculosis vaccine induces respiratory-mucosal immunity in humans. JCI Insight. 2022 Feb 8;7(3):e155655. doi: 10.1172/jci.insight.155655. PMID 34990408
- See also: Safety and immunopotency of an adenovirus-vectored tuberculosis vaccine delivered via inhaled aerosol to healthy humans: a dose and route comparison phase 1b study — https://www.medrxiv.org/content/10.1101/2021.09.09.21263339v1